CLINICAL TRIAL: NCT00038103
Title: Open-Label, Multicentre, Controlled Study Of Exemestane (Aromasin®) With Or Without Celecoxib (Celebrex®) In Postmenopausal Women With Advanced Breast Cancer (ABC) Having Progressed On Tamoxifen
Brief Title: Open-Label Study Of Exemestane With Or Without Celecoxib In Postmenopausal Women With ABC Having Progressed On Tamoxifen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NQ8-01-02-013; A3191139
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Active Comparator)
  Interventions: Drug: Exemestane
- 2. (Experimental)
  Interventions: Drug: Celecoxib + Exemestane

INTERVENTIONS:
Drug: Exemestane — Patient will be instructed to take a 25 mg exemestane tablet, once a day, every day, with food.
  Other Names: Aromasin
  Arms: 1.
Drug: Celecoxib + Exemestane — Exemestane + celecoxib treatment arm, she will be instructed to take also two x 200 mg celecoxib capsules twice a day, every day, with food.
  Other Names: Celebrex, Aromasin
  Arms: 2.

SUMMARY:
This is an open-label, multicenter, randomized (1:1 randomization ratio) study of either exemestane or exemestane plus celecoxib in postmenopausal women with ABC having progressed on tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female patient with histologically or cytologically confirmed breast cancer having progressed on Tamoxifen.
* Advanced disease: patients with advanced breast carcinoma with disease progression who had progressed/relapsed following > 8 weeks of treatment with Tamoxifen for advanced disease; or progressed during adjuvant Tamoxifen for at least 6 or 12 months depending on receptor status; or progressed within 12 months from completion of adjuvant treatment with Tamoxifen.
* at least one measurable lesion

Exclusion Criteria:

* More than one previous chemotherapy and/or more than one hormonotherapy for advanced disease.
* Previous hormonotherapy for advanced disease other than Tamoxifen.
* Myocardial infarction within previous 6 mo

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2002-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Pfizer Investigational Site, Dallas, Texas, United States
- Belgium (5):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Namur
  - Pfizer Investigational Site, Wilrijk
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Sydney, Nova Scotia, Canada
- Colombia (2):
  - Pfizer Investigational Site, Bogotá, Bogota . DC
  - Pfizer Investigational Site, Cali
- India (4):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
- Mexico (2):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Pfizer Investigational Site, Manila, Philippines

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NQ8-01-02-013&StudyName=Open-Label%20Study%20Of%20Exemestane%20With%20Or%20Without%20Celecoxib%20In%20Postmenopausal%20Women%20With%20ABC%20Having%20Progressed%20On%20Tamoxifen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects in the exemestane arm were never treated. One subject refused to be treated having originally consented to participate in this study and the other, reason for not starting treatment was unknown
Groups:
- Exemestane (Exemestane Alone): oral dose exemestane taken with food (25 mg tablet once daily)
- Combination (Exemestane + Celecoxib): oral doses to be taken with food (25 mg tablet exemestane once daily; celecoxib 2 x 200 mg tablets twice daily)
Period: Overall Study
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Started | 55 | 56
End of Treatment | 53 (patients remained on treatment until discontinued) | 56 (patients remained on treatment until discontinued)
Completed | 0 | 0
Not Completed | 55 | 56
Not completed — Adverse Event | 5 | 6
Not completed — Lack of Efficacy | 48 | 41
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Sponsor Decision | 0 | 1
Not completed — Randomized/never treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib) | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Customized [Number; unit: Participants]
  < 50 years | 20.0 | 16.0 | 36.0
  50-64 years | 20.0 | 27.0 | 47.0
  65-79 years | 15.0 | 12.0 | 27.0
  => 80 years | 0.0 | 1.0 | 1.0
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were female
  Participants
    Female | 55 | 56 | 111.0
    Male | 0 | 0 | 0.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinical Benefit
Description: Clinical benefit was based on objective tumor assessments made according to Response Evaluation Criteria (RECIST) system of unidimensional evaluation. Includes subjects with complete response (CR), partial response (PR), and long term disease stabilization (SD) for at least 24 weeks.
Time Frame: Baseline, Week 8, 16, 24, and every 12 weeks beyond 24 up to Week 108 and every 24 weeks thereafter until 9 months following last subject last visit (LSLV)
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 49 | 51
participants | 24 | 24
Statistical Analysis 1: Comparison: Exemestane (Exemestane Alone); Test type: Superiority or Other; Clinical Benefit Rate = 49.0, 95% CI [34.4 to 63.7] — Number of subjects showing clinical benefits out of the number of subjects in the evaluable set
Statistical Analysis 2: Comparison: Combination (Exemestane + Celecoxib); Test type: Superiority or Other; Clinical Benefit Rate = 47.1, 95% CI [32.9 to 61.5] — Number of subjects showing clinical benefits out of the number of subjects in the evaluable set

2. Secondary Outcome: Number of Subjects With Objective Response
Description: Objective tumor response includes subjects with CR or PR according to RECIST.
Time Frame: Baseline, Weeks 8, 16, 24, every 12 weeks from Week 24 up to Week 108, and every 24 weeks thereafter until 9 months following LSLV
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 49 | 51
participants | 11 | 12
Statistical Analysis 1: Comparison: Exemestane (Exemestane Alone); Test type: Superiority or Other; Objective Response Rate = 22.4, 95% CI [11.8 to 36.6] — Number of subjects showing objective response out of the number of subjects in the evaluable set
Statistical Analysis 2: Comparison: Combination (Exemestane + Celecoxib); Test type: Superiority or Other; Objective Response Rate = 23.5, 95% CI [12.8 to 37.5] — Number of subjects showing objective response out of the number of subjects in the evaluable set

3. Secondary Outcome: Duration of Clinical Benefit
Description: Time from randomization date to first objective documentation of tumor progression or death due to tumor progression in the absence of previous documentation of tumor progression.
Time Frame: as for outcome 2
Population: Evaluable population. Number of participants analyzed = number of subjects with clinical benefit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 24 | 24
weeks | 49.1 [37.0 to 85.0] | 96.6 [37.0 to 147.0]

4. Secondary Outcome: Duration of Objective Response (in Subjects With CR or PR)
Description: Time from the first objective documentation of response until the first objective documentation of tumor progression.
Time Frame: Baseline, Weeks 8, 16, 24, every 12 weeks beyond 24 up to Week 108, and every 24 weeks thereafter until 9 months following LSLV
Population: Evaluable population. Number of participants analyzed = number of subjects with objective response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 11 | 12
weeks | 32.7 [23.1 to 68.9] | 40.1 [28.3 to 169.1]

5. Secondary Outcome: Duration of Long-Term SD
Description: Time from start of treatment until the first objective documentation of tumor progression or death due to tumor progression in the absence of previous documentation of tumor progression in subjects with long-term SD.
Time Frame: Baseline, Weeks 8, 16, 24, every 12 weeks from Week 24 up to Week 108, and every 24 weeks thereafter until 9 months LSLV
Population: Evaluable population. Number of participants analyzed = number of subjects with long-term SD.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 13 | 12
weeks | 52.9 [36.6 to 110.0] | 109.7 [36.6 to 147.0]

6. Secondary Outcome: Time to Tumor Progression
Description: Time from randomization to first objective tumor recurrence or progression or death due to tumor progression in the absence of previous documentation of tumor progression.
Time Frame: Baseline, Weeks 8, 16, 24, every 12 weeks beyond Week 24 up to Week 108 and every 24 weeks thereafter until 9 months following LSLV
Population: Evaluable population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 49 | 51
weeks | 20 [9.4 to 36.6] | 23.4 [16.3 to 36.9]

7. Secondary Outcome: Time to Treatment Failure
Description: Time from randomization to first objective tumor recurrence or progression or death due to any cause or withdrawal from study treatment due to any reason, whichever was the earliest.
Time Frame: as for outcome 2
Population: Evaluable population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 49 | 51
Weeks | 18.1 [9.3 to 36.6] | 20.4 [14.9 to 34.6]

8. Secondary Outcome: Survival
Description: Time from randomization to date of death (any cause).
Time Frame: Baseline, Weeks 8, 16, 24, every 12 weeks from Week 24 up to Week 108, and every 24 weeks thereafter until 9 months following LSLV or death
Population: Evaluable population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Number analyzed (Participants) | 49 | 51
weeks | 74.4 [57.7 to 101.4] | 73.9 [52.3 to 106.7]

ADVERSE EVENTS:
Arm/Group | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Serious Adverse Events (participants affected / at risk) | 9 | 14
Other Adverse Events (participants affected / at risk) | 45 | 43
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Jaundice (Hepatobiliary disorders) | 2/53 | 0/56
Pain (General disorders) | 1/53 | 1/56
Post procedural complication (Reproductive system and breast disorders) | 1/53 | 0/56
Death (General disorders) | 1/53 | 1/56
Ascites (Gastrointestinal disorders) | 1/53 | 0/56
Nausea (Gastrointestinal disorders) | 1/53 | 0/56
Vomiting (Gastrointestinal disorders) | 2/53 | 0/56
General physical health deterioration (General disorders) | 1/53 | 1/56
Asterixis (Nervous system disorders) | 1/53 | 0/56
Deep Vein Thrombosis (Vascular disorders) | 1/53 | 1/56
Neck Pain (Musculoskeletal and connective tissue disorders) | 1/53 | 0/56
Gait Disturbance (General disorders) | 1/53 | 1/56
Disorientation (Psychiatric disorders) | 1/53 | 0/56
Asthenia (General disorders) | 2/53 | 0/56
Dizziness (Psychiatric disorders) | 1/53 | 0/56
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/56
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/53 | 3/56
Cough (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/56
Intestinal Obstruction (Gastrointestinal disorders) | 1/53 | 0/56
Knee Arthroplasty (Surgical and medical procedures) | 0/53 | 1/56
Scleroderma (Musculoskeletal and connective tissue disorders) | 0/53 | 1/56
Miller Fisher Syndrome (Nervous system disorders) | 0/53 | 1/56
Polyneuropathy (Nervous system disorders) | 0/53 | 1/56
Diarrhoea (Gastrointestinal disorders) | 0/53 | 1/56
Fatigue (General disorders) | 0/53 | 1/56
Paresis (Nervous system disorders) | 0/53 | 1/56
Fall (Injury, poisoning and procedural complications) | 0/53 | 1/56
Back Pain (General disorders) | 0/53 | 1/56
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0/53 | 1/56
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 | 1/56
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0/53 | 1/56
Cardiac Failure Congestive (Cardiac disorders) | 0/53 | 1/56
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 0/53 | 1/56
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 | 1/56
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exemestane (Exemestane Alone) | Combination (Exemestane + Celecoxib)
Tinnitus (Ear and labyrinth disorders) | 1/53 | 0/53
Vertigo (Ear and labyrinth disorders) | 1/53 | 1/53
Conjunctivitis (Eye disorders) | 1/53 | 0/53
Abdominal pain (Gastrointestinal disorders) | 2/53 | 3/53
Abdominal pain upper (Gastrointestinal disorders) | 2/53 | 3/53
Ascites (Gastrointestinal disorders) | 1/53 | 0/53
Cheilitis (Gastrointestinal disorders) | 1/53 | 0/53
Constipation (Gastrointestinal disorders) | 4/53 | 0/53
Diarrhoea (Gastrointestinal disorders) | 3/53 | 5/53
Dysphagia (Gastrointestinal disorders) | 1/53 | 0/53
Faecal incontinence (Gastrointestinal disorders) | 1/53 | 1/53
Gastritis (Gastrointestinal disorders) | 1/53 | 2/53
Intestinal obstruction (Gastrointestinal disorders) | 1/53 | 0/53
Nausea (Gastrointestinal disorders) | 5/53 | 3/53
Odynophagia (Gastrointestinal disorders) | 1/53 | 0/53
Oesophagitis (Gastrointestinal disorders) | 1/53 | 0/53
Peptic ulcer (Gastrointestinal disorders) | 1/53 | 0/53
Toothache (Gastrointestinal disorders) | 1/53 | 0/53
Vomiting (Gastrointestinal disorders) | 8/53 | 2/53
Asthenia (General disorders) | 4/53 | 6/53
Axillary pain (General disorders) | 1/53 | 0/53
Chest pain (General disorders) | 2/53 | 2/53
Death (General disorders) | 1/53 | 0/53
Fatigue (General disorders) | 4/53 | 3/53
Gait disturbance (General disorders) | 2/53 | 2/53
General physical health deterioration (General disorders) | 1/53 | 1/53
Inflammation (General disorders) | 1/53 | 0/53
Oedema (General disorders) | 1/53 | 0/53
Oedema peripheral (General disorders) | 2/53 | 2/53
Pain (General disorders) | 2/53 | 2/53
Pyrexia (General disorders) | 1/53 | 0/53
Ulcer haemorrhage (General disorders) | 1/53 | 0/53
Jaundice (Hepatobiliary disorders) | 2/53 | 1/53
Hypersensitivity (Immune system disorders) | 1/53 | 0/53
Fungal infection (Infections and infestations) | 1/53 | 0/53
Gastroenteritis (Infections and infestations) | 1/53 | 0/53
Lymphangitis (Infections and infestations) | 1/53 | 0/53
Respiratory tract infection (Infections and infestations) | 2/53 | 0/53
Sinusitis (Infections and infestations) | 1/53 | 1/53
Upper respiratory tract infection (Infections and infestations) | 1/53 | 1/53
Urinary tract infection (Infections and infestations) | 1/53 | 5/53
Fall (Injury, poisoning and procedural complications) | 1/53 | 1/53
Joint dislocation (Injury, poisoning and procedural complications) | 1/53 | 0/53
Medical device complication (Injury, poisoning and procedural complications) | 1/53 | 0/53
Post procedural complication (Injury, poisoning and procedural complications) | 1/53 | 0/53
Wound (Injury, poisoning and procedural complications) | 1/53 | 0/53
Alanine aminotransferase increased (Investigations) | 1/53 | 1/53
Aspartate aminotransferase (Investigations) | 1/53 | 1/53
Blood alkaline phosphatase (Investigations) | 2/53 | 0/53
Blood alkaline phosphatase increased (Investigations) | 2/53 | 0/53
Gamma-glutamyltransferase (Investigations) | 1/53 | 1/53
Low density lipoprotein (Investigations) | 1/53 | 0/53
Neutrophil count decreased (Investigations) | 1/53 | 0/53
Platelet count decreased (Investigations) | 1/53 | 0/53
Weight decreased (Investigations) | 2/53 | 1/53
Weight increased (Investigations) | 2/53 | 0/53
White blood cell count decreased (Investigations) | 1/53 | 0/53
Anorexia (Metabolism and nutrition disorders) | 7/53 | 3/53
Diabetes mellitus (Metabolism and nutrition disorders) | 1/53 | 0/53
Hypercalcaemia (Metabolism and nutrition disorders) | 1/53 | 0/53
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2/53 | 0/53
Hyperglycaemia (Metabolism and nutrition disorders) | 3/53 | 1/53
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2/53 | 0/53
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1/53 | 0/53
Hypocalcaemia (Metabolism and nutrition disorders) | 4/53 | 0/53
Hypoglycaemia (Metabolism and nutrition disorders) | 1/53 | 0/53
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/53 | 6/53
Back pain (Musculoskeletal and connective tissue disorders) | 8/53 | 10/53
Bone pain (Musculoskeletal and connective tissue disorders) | 2/53 | 5/53
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1/53 | 0/53
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/53 | 0/53
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/53 | 2/53
Myalgia (Musculoskeletal and connective tissue disorders) | 3/53 | 2/53
Neck pain (Musculoskeletal and connective tissue disorders) | 1/53 | 1/53
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7/53 | 5/53
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/53 | 0/53
Asterixis (Nervous system disorders) | 1/53 | 0/53
Ataxia (Nervous system disorders) | 1/53 | 0/53
Dizziness (Nervous system disorders) | 2/53 | 0/53
Headache (Nervous system disorders) | 5/53 | 4/53
Hypoaesthesia (Nervous system disorders) | 1/53 | 1/53
Paraesthesia (Nervous system disorders) | 2/53 | 2/53
Peripheral sensory neuropathy (Nervous system disorders) | 1/53 | 3/53
Peroneal nerve palsy (Nervous system disorders) | 1/53 | 0/53
Sensory loss (Nervous system disorders) | 1/53 | 0/53
Anxiety (Psychiatric disorders) | 1/53 | 0/53
Confusional state (Psychiatric disorders) | 1/53 | 0/53
Disorientation (Psychiatric disorders) | 1/53 | 0/53
Insomnia (Psychiatric disorders) | 3/53 | 1/53
Dysuria (Renal and urinary disorders) | 2/53 | 0/53
Proteinuria (Renal and urinary disorders) | 3/53 | 0/53
Pyuria (Renal and urinary disorders) | 1/53 | 0/53
Urinary incontinence (Renal and urinary disorders) | 1/53 | 0/53
Breast pain (Reproductive system and breast disorders) | 1/53 | 2/53
Pelvic pain (Reproductive system and breast disorders) | 1/53 | 1/53
Vaginal discharge (Reproductive system and breast disorders) | 1/53 | 0/53
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/53 | 0/53
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/53 | 0/53
Cough (Respiratory, thoracic and mediastinal disorders) | 9/53 | 4/53
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2/53 | 0/53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4/53 | 7/53
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2/53 | 0/53
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/53
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/53
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/53 | 1/53
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/53
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/53
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1/53 | 0/53
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2/53 | 1/53
Pruritus (Skin and subcutaneous tissue disorders) | 3/53 | 0/53
Rash (Skin and subcutaneous tissue disorders) | 3/53 | 2/53
Deep vein thrombosis (Vascular disorders) | 1/53 | 1/53
Hot flush (Vascular disorders) | 6/53 | 8/53
Hypertension (Vascular disorders) | 1/53 | 2/53
Lymphoedema (Vascular disorders) | 1/53 | 0/53
Pallor (Vascular disorders) | 1/53 | 1/53
Phlebitis (Vascular disorders) | 1/53 | 0/53
Vasodilatation (Vascular disorders) | 1/53 | 0/53
Anaemia (Blood and lymphatic system disorders) | 0/53 | 2/53
Cardiac failure congestive (Cardiac disorders) | 0/53 | 1/53
Visual impairment (Eye disorders) | 0/53 | 1/53
Abdominal discomfort (Gastrointestinal disorders) | 0/53 | 1/53
Gastrointestinal pain (Gastrointestinal disorders) | 0/53 | 1/53
Mouth ulceration (Gastrointestinal disorders) | 0/53 | 1/53
Malaise (General disorders) | 0/53 | 1/53
Acarodermatitis (Infections and infestations) | 0/53 | 1/53
Breast cellulitis (Infections and infestations) | 0/53 | 1/53
Bronchitis (Infections and infestations) | 0/53 | 3/53
Bronchitis viral (Infections and infestations) | 0/53 | 1/53
Ear infection (Infections and infestations) | 0/53 | 1/53
Influenza (Infections and infestations) | 0/53 | 2/53
Nasopharyngitis (Infections and infestations) | 0/53 | 2/53
Tinea pedis (Infections and infestations) | 0/53 | 1/53
Tooth infection (Infections and infestations) | 0/53 | 1/53
Tracheitis (Infections and infestations) | 0/53 | 1/53
Wrist fracture (Injury, poisoning and procedural complications) | 0/53 | 1/53
Alanine aminotransferase (Investigations) | 0/53 | 1/53
Hepatic enzyme increased (Investigations) | 0/53 | 1/53
Pulse pressure increased (Investigations) | 0/53 | 1/53
Hypoproteinaemia (Metabolism and nutrition disorders) | 0/53 | 1/53
Flank pain (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/53 | 2/53
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Scleroderma (Musculoskeletal and connective tissue disorders) | 0/53 | 1/53
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 | 1/53
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 | 1/53
Brachial plexopathy (Nervous system disorders) | 0/53 | 1/53
Carpal tunnel syndrome (Nervous system disorders) | 0/53 | 1/53
Dysaesthesia (Nervous system disorders) | 0/53 | 1/53
Dysarthria (Nervous system disorders) | 0/53 | 1/53
Miller Fisher syndrome (Nervous system disorders) | 0/53 | 1/53
Paresis (Nervous system disorders) | 0/53 | 1/53
Polyneuropathy (Nervous system disorders) | 0/53 | 1/53
Somnolence (Nervous system disorders) | 0/53 | 2/53
Urge incontinence (Renal and urinary disorders) | 0/53 | 1/53
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/53 | 1/53
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/53 | 1/53
Alopecia (Skin and subcutaneous tissue disorders) | 0/53 | 2/53
Dermatitis (Skin and subcutaneous tissue disorders) | 0/53 | 1/53
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/53 | 1/53
Eczema (Skin and subcutaneous tissue disorders) | 0/53 | 1/53
Skin lesion (Skin and subcutaneous tissue disorders) | 0/53 | 1/53
Cholecystectomy (Surgical and medical procedures) | 0/53 | 1/53
Knee arthroplasty (Surgical and medical procedures) | 0/53 | 1/53
Hypotension (Vascular disorders) | 0/53 | 1/53
Varicose vein (Vascular disorders) | 0/53 | 1/53
Dyspepsia (Gastrointestinal disorders) | 0/53 | 2/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.